CLINICAL TRIAL: NCT04642690
Title: The Association Between Nitrates, Nitrosylated Proteins, and Interleukin-8 in Barrett's Esophagus and Esophageal Adenocarcinoma
Brief Title: Nitrates and IL-8 in Barrett's Esophagus
Status: Terminated | Type: Observational
Why Stopped: could not collect adequate samples
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cadman Leggett, Principal Investigator, Mayo Clinic
Other Study IDs: 20-004618
Record Dates: First submitted 2020-10-09; First posted 2020-11-24 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Group 1-NSE: Patients found to have grossly normal squamous epithelium during endoscopy
- Group 2-EEG: Patients found to have grossly apparent erosive esophagitis >1cm with Los Angeles Classification A-D
- Group 3-NDBE Short: Patients with non-dysplastic Barrett's Esophagus (NDBE) > 1cm (Short Segment)
- Group 4-NDBE Long: Patients with non-dysplastic Barrett's Esophagus (NDBE) > 1cm (Long Segment)
- Group 5: Barrett's Esophagus (BE) with high-grade dysplasia (HGD) or esophageal adenocarcinoma (EAC)
- Group 6-Esophagectomy: Patients undergoing resection of esophageal cancer
- Group -7 Pilot and Feasibility: Patients undergoing EGD with NSE, NDBE, BE-HGD, or EAC for feasibility of analytical techniques

SUMMARY:
The purpose of this study is to determine if nitrates and IL-8 (which are found in food and throughout the body regulating stomach acidity) play a role in Barrett's Esophagus and/or Esophageal Adenocarcinoma severity and if screening for these biomarkers can help predict patients that are more at risk for developing worsening disease.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing a clinicallly-indicated Esophagogastroduoedoscopy (EGD).

Exclusion Criteria:

* Comorbid inflammatory medical condition.
* Use of antiinflammatory (aspirin and NSAIDs) or immunosuppressants over the past 1 week.
* Use of nitrate containing medication in the past 1 week.
* Consumption of nitrate rich foods in preceding 24 hours.
* Known allergy to meat or nitrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult individuals scheduled for clinically indicated EGD procedure. Subjects with normal squamous epithelium, erosive esophagitis, or varying degrees of Barrett's Esophagus may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Nitrate Levels | Baseline
  Nitrate levels in serum, saliva and tissue in patients with normal squamous epithelium, erosive esophagitis, non-dysplastic BE (NDBE), and BE with high-grade dysplasia (HGD) or EAC
Serum and Tissue Biomarkers | Baseline
  Levels of IL-8 in patients diagnosed BE dysplasia and EAC

SECONDARY OUTCOMES:
Biomarkers and disease progression | Baseline
  Level of IL-8 in serum and tissue in patients with NDBE that progressed to BE

CONTACTS AND LOCATIONS:
Overall Officials: Cadman Leggett, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No